CLINICAL TRIAL: NCT03614624
Title: Left Ventricular 2D and 3D Strain in Healthy Subject : Comparative Study Between Two Echocardiograph (Vivid 9 General Electric et Epiq 7 Philips)
Brief Title: Study C3S : Comparison Among Healthy Subject
Acronym: RBHPCLERFOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-402; 2016-A01584-47 (Other: 2016-A01584-47)
Record Dates: First submitted 2018-07-20; First posted 2018-08-03 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy subject; Echocardiography; 2D and 3D Strain; General Electric; Philips

STUDY DESIGN:
Intervention Model Description: All the healthy volunteers who consent to participate in the study, and who are eligible according to the protocol will have an clinical examination, an electrocardiogram and an echocardiography with two devices.
Masking Description: No masking description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of two devices (Experimental): Patients receive clinical examination, electrocardiogramm and echocardiography.
  Interventions: Device: Comparative standard echocardiography between two devices : Vivid 9 General Electric and Epiq 7 Philips

INTERVENTIONS:
Device: Comparative standard echocardiography between two devices : Vivid 9 General Electric and Epiq 7 Philips — Comparison of the various values of strain with the echograph General Electric and the electrograph Philips.

SUMMARY:
The aim of the C3S study is research an equivalence with longitudinal, radial and circumferential, global and segmental strain value, in left Ventricular in 2 and 3 dimension between two echograph General Electric Vivid 9 (GE Vingmed, Horton, Norway) et Philips Epiq 7.

DETAILED DESCRIPTION:
Healthy volunteer will be inform about the study by email and press. They could join the clinical research team by email and phone to ask more questions about the study. Then the investigator, verify the eligibiliy of the volunteers and schedule an appointment for the visit of inclusion. During this visit, the patient's consent will be collected. One echocardiography will be complete on echograph General Electric Vivid 9 to collect the clinical data necessary for the study and to eliminate the presence of criteria of exclusions, the acquisition of the loops of ultrasound will be realized on both echographs by a first investigator. A second investigator will make the post-treatment of the ultrasound images on consoles ECHOPAC PC version 201, General Electric Medical System and Q Station version 3.5, Philips Healthcare in two different times, to obtain the values of the various strain.

Furthermore, an clinical exam, an ECG, a questionnary will be realized.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years' old
* Without any cardiac pathology
* Not taking long-term treatments, except oral contraception
* Consented to participate in the study

Exclusion Criteria:

* Existence of heart disease : myocardial revascularization, primitive cardiopathy (dilated or hypertrophic cardiopathy), moderate or severe valvulopathy, pulmonary hypertension, congenital heart disease operated or not, previous cardiac heart failure, previous rhythm disturbance and/or pacemaker, hypertension treated or untreated, peripheral artery disease : occlusive arteriopathy of the lower limbs, peripheral arterial aneurysm, stenosis or peripheral arterial occlusion.
* Practicing intensive sport (more than 6 hours per week)
* Untreated type 2 or 1 diabetes , treated dyslipidemia, chronic alcoholic intoxication (men more than 3 units of alcohol per day and women more than 2 units per day)
* Existence of heart disease or previous heart disease
* Pregnant or lactating women,
* Dependent adult
* Patients minor,
* Decline the study,
* Existence of a psychiatric pathology
* Inability to grant its informed consent
* No affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Value of the longitudinal strain value, in left Ventricular in 2 and 3 dimension. | 1 year
  The acquisition of the ultrasound loops on both echographs is realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.
Values of the radial strain value, in left Ventricular in 2 and 3 dimension. | 1 year
  The acquisition of the ultrasound loops on both echographs is realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.
Values of the circumferential strain value, in left Ventricular in 2 and 3 dimension. | 1 year
  The acquisition of the ultrasound loops on both echographs is realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.
Values of the global strain value, in left Ventricular in 2 and 3 | 1 year
  The acquisition of the ultrasound loops on both echographs is realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.
Values of the segmental strain value, in left Ventricular in 2 and 3 | 1 year
  The acquisition of the ultrasound loops on both echographs is realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.

SECONDARY OUTCOMES:
Values of longitudinal global strain of the right ventricle between two echographs (General Electric and Philips). | 1 year
  The acquisition of the ultrasound loops on both echographs are realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.
Values of segmental 2D of the right ventricle between two echographs (General Electric and Philips). | 1 year
  The acquisition of the ultrasound loops on both echographs are realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.
Values of strain 2D of the left atrium between two echographs (General Electric and Philips). | 1 year
  The acquisition of the ultrasound loops on both echographs are realized at the same time. The various values of strain are obtained after post-treatment of the ultrasound loops on ECHOPAC PC version 201 software for the echograph General Electric and the Q Station version 3.5 software for the echograph Phillips. The post-treatment on both software are made in two different times to avoid possible biases.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CLERFOND, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France